CLINICAL TRIAL: NCT00718783
Title: Molecular Analysis of Retinoblastoma
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MARB; 1R01EY018599 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Each tumor sample will be immediately transferred to a sterile cryovial and flash frozen in liquid nitrogen.
  * White blood cells will be isolated from the blood sample as a source of genomic DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retinoblastoma
  Interventions: Other: Tissue samples taken from retinoblastoma; Other: 5 ml peripheral blood

INTERVENTIONS:
Other: Tissue samples taken from retinoblastoma — Tissue banking
Other: 5 ml peripheral blood — White blood cells will be isolated from the blood sample as a source of genomic DNA.

SUMMARY:
Retinoblastoma is a childhood tumor of the retina that affects approximately 1 in 18,000 children. Retinoblastoma is more prevalent in Central America, where most patients present with advanced intraocular and extraocular disease. Therefore, we have formed collaboration with Central American investigators to provide us with frozen retinoblastoma tumors from patients undergoing routine enucleation. The objective of this protocol is to begin to identify the mutations and gene expression changes that occur in retinoblastoma cells following RB1 gene inactivation in order to more effectively target chemotherapy for treating bilateral retinoblastoma.

DETAILED DESCRIPTION:
This is a biology protocol with no treatment regimen associated. Following routine enucleation of the retinoblastoma affected eye, a portion of the tumor will be removed and flash frozen and sent to St. Jude for RNA and DNA analysis. Some tissue will undergo histopathological analysis and tissue microarrays will be isolated.

ELIGIBILITY:
Inclusion Criteria:

* Must have clinical diagnosis of retinoblastoma (to be confirmed histologically after enucleation)
* Legal guardians must willing to sign an informed consent indicating that they are aware of this study and its possible benefits. Legal guardians will be given a copy of the consent form.
* Patient is being seen at this AHOPCA institution:

Exclusion Criteria:

* Ophthalmologist or oncologist is concerned that sampling will interfere with staging.
* Diagnosis other than retinoblastoma.
* Affiliated hospital is unable to provide pathologic evidence of retinoblastoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Identify genes exhibiting differential expression within intraocular disease tissue between patients having only intraocular involvement and those having extraocular involvement. | Indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Brennan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- Hospital Calvo Mackenna, Santiago, Santiago Metropolitan, Chile
- Hospital Escuela Bloque Materno Infantil, Tegucigalpa, Honduras

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols